CLINICAL TRIAL: NCT02978989
Title: A Randomized Controlled Trial Comparing a Solo and Non-solo Approach for Laparoscopic Cholecystectomy
Brief Title: Solo and Non-solo Approach for Laparoscopic Cholecystectomy
Acronym: SOLOGB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daejeon St. Mary's hospital (Other)
Responsible Party: Principal Investigator, Say-June Kim, Professor, Daejeon St. Mary's hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SSGB-1
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Cholecystectomy, Laparoscopic
Keywords: Laparoscopic cholecystectomy; Solo surgery; Camera holder; Cholecystitis
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LC & nonsolo approach (Placebo Comparator): The surgical intervention is nonsolo LC.
  Interventions: Procedure: nonsolo LC
- LC & solo approach (Active Comparator): The surgical intervention is solo LC.
  Interventions: Procedure: solo LC

INTERVENTIONS:
Procedure: nonsolo LC — This patient is scheduled to undergo nonsolo laparoscpic cholecystectomy.
  Other Names: Nonsolo laparoscopic cholecystectomy
  Arms: LC & nonsolo approach
Procedure: solo LC — This patient is scheduled to undergo solo laparoscpic cholecystectomy.
  Other Names: Solo laparoscopic cholecystectomy
  Arms: LC & solo approach

SUMMARY:
To determine the safety and feasibility of solo laparoscopic cholecystectomy, which is defined as the application of solo surgery to laparoscopic cholecystectomy, by comparing consecutive non-solo procedures conducted by a surgeon in the presence or absence of human assistant(s).

DETAILED DESCRIPTION:
Laporoscopic cholecystectomy usually requires three surgeons, including an operator, a camera assistant, and other instrument assistant. Recent advancement of technology made it possible to develop the conveniently adjustable holders for camera and other laparoscopic instruments. The application of these instruments enables "solo-surgery" wherein an operation is driven by single surgeon. During surgery, human assistant(s) are helpful because of their instant assistance according to the operation's need. Therefore, the utilization of instruments instead of human assistants would be cumbersome. However, the utilization of instruments would be helpful by enabling operation-driven repositioning of the camera and instrument(s). Currently, no attempt has been made to objectively compare the merits and demerits of these two procedures. Therefore, this study was conducted to determine the safety and feasibility of solo laparoscopic cholecystectomy, which is defined as the application of solo surgery to laparoscopic cholecystectomy, by comparing consecutive non-solo procedures conducted by a surgeon in the presence or absence of human assistant(s).

ELIGIBILITY:
Inclusion Criteria:

1. The patients planed to undergo elective laparoscopic cholecystectomy
2. Benign gallbladder diseases requiring surgery
3. The patients who are indicated for single-port laparoscopic cholecystectomy.

Exclusion Criteria:

1. the patients with complicated cholecystitis
2. the patients with the gallbladder with a thickness more than 4mm.
3. the patients who are expected to have severe peritoneal adhesion.
4. the patients with malignant gallbladder diseases.
5. the patients whose operation appears to need human assistant(s)

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Operation time | day 1
  Operation time correlates with surgical difficulity.

SECONDARY OUTCOMES:
Pain score | day 3
  Daily pain scores are assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Say-June Kim, M.D., Ph.D., Principal Investigator — Daejeon St. Mary's hospital, the Catholic University of Korea, 222, Banpo-dong, Seocho-gu, Seoul, 06591, South Korea

IPD SHARING:
Plan to Share IPD: No